CLINICAL TRIAL: NCT03997825
Title: Five-Plus Year Follow-Up of SMART (Surgical Multicenter Assessment of RF Ablation for the Treatment of Vertebrogenic Back Pain) Trial
Brief Title: Five-Plus Year Follow-Up of SMART Randomized Controlled Trial
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Relievant Medsystems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP 0011
Record Dates: First submitted 2019-05-07; First posted 2019-06-25 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Basivertebral Nerve (BVN) Ablation — Single follow-up visit of previously treated participants from the SMART trial.

SUMMARY:
The objective of this study is to evaluate long-term ongoing effectiveness of the Intracept Intraosseous Nerve Ablation System for the treatment of chronic low back pain.

DETAILED DESCRIPTION:
This is a prospective multi-center, nonintervention, observational, single arm post market data collection of the 5+ year effectiveness and satisfaction outcome for the SMART trial population.

ELIGIBILITY:
Inclusion Criteria:

* LBP at least 6 months from original SMART Trial
* RF Ablation Arm from SMART Trial

Exclusion Criteria:

-Control Arm Subjects from SMART Trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 117 U.S. subjects treated per protocol in the treatment arm of the original SMART trial in the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Fischgrund, MD, Principal Investigator — Corewell Health East
Locations (13):
- United States (13):
  - Desert Institute for Spine Care, Phoenix, Arizona
  - SpineCare Medical Group, Daly City, California
  - Memorial Orthopedic Surgical Group, Long Beach, California
  - Cedars Sinai Spine Center, Los Angeles, California
  - Drug Studies of America, Marietta, Georgia
  - Indiana Spine Group, Carmel, Indiana
  - Maine Medical Partners, Scarborough, Maine
  - Michigan Orthopedics Instititute, Southfield, Michigan
  - OrthoCarolina, Charlotte, North Carolina
  - Pacific Sports and Spine, Eugene, Oregon
  - Rothman Orthopedic Institute, Bensalem, Pennsylvania
  - Seton Spine and Scoliosis Center, Austin, Texas
  - Virginia iSpine Physicians, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- BVN Ablation Arm: Per protocol successfully treated United States participants randomized to BVN Ablation arm in the original SMART RCT
Period: Overall Study
Arm/Group | BVN Ablation Arm
Started | 117
Completed | 100
Not Completed | 17
Not completed — Death | 3
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 3
Not completed — Refused participation | 1

BASELINE CHARACTERISTICS:
Groups:
- BVN Ablation Arm: Randomized and successfully treated with basivertebral nerve ablation
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 94
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Baseline Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — The Oswestry Disability Index (ODI) is a validated questionnaire of low back pain-related disability (impact of low back pain on function) with a scale of 0 to 100. It is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be 10-12 points for minimally invasive procedures.
  units on a scale | 42.8 (11.6)
Baseline Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The VAS pain questionnaire involves a 10 cm scale scale with 0 being no pain and 10 being worst imaginable pain. Participants are asked to indicate on the scale the degree of pain as an average level of low back pain for the last 7 days. Literature reports a minimally clinically important difference in VAS of 1.5 to 2.0 cm/point difference.
  units on a scale | 6.73 (1.43)

OUTCOME MEASURES:

1. Primary Outcome: LS Mean Reduction in Oswestry Disability Index (ODI) From Baseline
Description: Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Difference in mean ODI at baseline and 5 years post treatment measurements.
Time Frame: Difference between baseline and 5 year post treatment measurements
Population: US per protocol BVN ablation treated participants who consented to participate
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale of 0 to 100 points
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
units on a scale of 0 to 100 points | 25.95 (18.54)
Statistical Analysis 1: Comparison: BVN Ablation Arm; Test type: Superiority; p = 0.001, ANCOVA

2. Secondary Outcome: LS Mean Reduction in VAS From Baseline
Description: Numeric pain scale with minimum of 0 to maximum of 10; with 0 being no pain and 10 being worst imaginable pain. Difference in mean VAS at baseline and at 5 years post treatment.
Time Frame: Difference between baseline and 5 year post treatment measurements
Population: US per protocol BVN ablation treated participants who consented to participate
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale of 0 to 10
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
score on a scale of 0 to 10 | 4.38 (2.35)
Statistical Analysis 1: Comparison: BVN Ablation Arm; Test type: Superiority; p = 0.001, ANCOVA

3. Secondary Outcome: Responder Rates
Description: Proportion of participants that achieve a threshold of > 15 point reduction in ODI and > 2 point reduction in VAS calculated as the difference between the baseline measurements and the 5 year post treatment measurements.
Time Frame: At 5 year post treatment
Population: US per protocol BVN ablation treated participants who consented to participate
Measure: Count of Participants; unit: Participants
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
Participants | 75

4. Secondary Outcome: Narcotics Use
Description: Proportion of participants using a narcotic more than once per week in the 30 days prior to the study visit. Difference in baseline to 5 year post treatment percentage measurements.
Time Frame: Difference between baseline and 5 years post treatment.
Population: US per protocol BVN ablation treated participants that consented to participate
Measure: Count of Participants; unit: Participants
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
Participants | 8

5. Secondary Outcome: Injections
Description: Proportion of participants receiving an injection for low back pain (adjudicated as same location and etiology as BVN ablation treatment) compared to baseline. Difference in percentage of participants at baseline and 5 years post treatment measurements.
Time Frame: Difference from baseline percentage measurement to 5 years post treatment measurement
Population: US per protocol BVN ablation treated participants that consented to participate
Measure: Count of Participants; unit: Participants
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
Participants | 1

6. Secondary Outcome: Interventions
Description: Proportion of participants receiving a pain intervention or surgery for low back pain (adjudicated as the same location and etiology as BVN ablation treatment) from procedure date to 5 year visit date.
Time Frame: Measured form treatment data to 5 years post treatment visit date
Population: US per protocol BVN ablation treated participants that consented to participate
Measure: Count of Participants; unit: Participants
Arm/Group | BVN Ablation Arm
Number analyzed (Participants) | 100
Participants | 11

ADVERSE EVENTS:
Time Frame: 5 years (mean of 6.4 years post BVN ablation)
Arm/Group | BVN Ablation Arm
All-Cause Mortality (participants affected / at risk) | 3/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03997825/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03997825/SAP_001.pdf